CLINICAL TRIAL: NCT03957551
Title: Cabozantinib and Pembrolizumab as a Front-line Therapy for Advanced Metastatic Melanoma
Brief Title: Cabozantinib and Pembrolizumab for Advanced Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to changes in the treatment of melanoma
Sponsor: John Rieth (Other)
Collaborators: Exelixis (Industry); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, John Rieth, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201904712
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Advanced Metastatic Melanoma
MeSH Terms: interventions — cabozantinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib and pembrolizumab (Experimental): Cabozantinib will be administered in the tablet form, at three dose levels: 40, 20 and 60 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Interventions: Drug: Cabozantinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form, at three dose levels: 40, 20 and 60 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Other Names: XL184; COMETRIQ™; Cabometyx®
Drug: Pembrolizumab — Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
  Other Names: Keytruda

SUMMARY:
The study aims to evaluate the safety and preliminary efficacy of the combination of cabozantinib and pembrolizumab in advanced melanoma

DETAILED DESCRIPTION:
This is an open-label, Phase 1b/2 trial for adults with advanced melanoma. The objective of the Phase 1b portion of the study is to establish the recommended Phase 2 dose of cabozantinib in combination with pembrolizumab in patients with unresectable melanoma and assess the safety and tolerability of the combined treatments. The objective of the Phase 2 portion of the study is to evaluate the preliminary efficacy of the established dose of cabozantinib in combination with pembrolizumab as measured by best overall response rate (ORR) (complete response [CR] + partial response [PR]) with the combination of agents in patients with unresectable stage III or stage IV melanoma.

ELIGIBILITY:
INCLUSION CRITERIA:

A patient must meet all of the following criteria to be eligible for enrollment (defined as receiving the first trial treatment) in the trial:

1. Histologically or cytologically confirmed unresectable in-transit (stage IIIc) or metastatic (stage IV) melanoma.
2. Must have at least 1 lesion that qualifies as a measurable (target) lesion per RECIST v1.1
3. Subjects must be willing to have blood draws for future biomarker testing as outlined in Section 11.9 of the protocol.
4. The subject has an ECOG performance score of </= 2 However; the phase 1b part will include only ECOG performance of 0-1 and life expectancy of >12 weeks
5. Aged 18 years and older.
6. The subject should not have received any treatment for advanced melanoma, EXCEPT, BRAF and/or MEK inhibitor. (2 week washout)
7. The subjects who have received adjuvant therapy including anti- PD-1 can be included in the study, if the last dose of the adjuvant treatment was >/= 6 months prior to developing metastatic relapse.
8. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
9. Female patients of childbearing potential, must have a negative urine or serum pregnancy test within 72 hours prior to taking the first dose of study medication, if.

   • If the urine test is positive or cannot be confirmed as negative then a serum test is required which must be negative for the patient to enroll.

   • Women of childbearing potential (WOCBP) must be willing to use 2 medically acceptable methods of contraceptive from Day 1 through 120 days after the last dose of trial treatment. The 2 medically acceptable birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide as per local regulations or guidelines. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
   * Male patients of reproductive potential must agree to use an adequate method of contraception from Day 1 through 120 days after the last dose of trial treatment. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
10. Able to swallow pills.
11. The subject must have recovered to baseline or < Grade 1 CTCAE v 4 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and /or stable on supportive therapy.

EXCLUSION CRITERIA:

A patient meeting any of the following criteria is not eligible to participate in this study:

1. Subject had prior treatment with any anti-PD-1, anti-PD-L1, or anti- PD-L2 agent for the treatment of advanced melanoma (although prior use in adjuvant setting is allowed if the last dose > 6 months prior developing metastatic disease).
2. Subjects with diagnosis of ocular and mucosal melanoma
3. Subject had prior cabozantinib for any indication.
4. Subject who received any small molecule tyrosine kinase inhibitor within 2 weeks before first dose of study treatment.
5. Subject who has had chemotherapy, radioactive, or biological cancer therapy within four weeks prior to the first dose of study drug, or who has not recovered to CTCAE Grade 1 or better from the AEs due to cancer therapeutics administered more than four weeks earlier.
6. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
7. Patient is currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of study drug. (A patient in the Survival Follow up phase of an investigational agent where no further treatment is expected is eligible).Patient is expected to require any other form of systemic or localized antineoplastic therapy while on study.
8. Patient is on any systemic corticosteroid therapy (more than 10 mg daily of prednisone or equivalent) within one week before the planned date for first dose of randomized treatment or on any other form of immunosuppressive medication.
9. Patient has a history of a malignancy (other than the disease under treatment in the study) within 2 years prior to first study drug administration. This should exclude adequately treated Stage 1 or Stage 2 basal/squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or other in situ cancers. Shorter intervals can be considered after discussion with Sponsor.
10. Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by MRI for at least four weeks prior to the first dose of study drug), have no evidence of new or enlarging brain metastases, neurologically asymptomatic and are off systemic steroids for at least two weeks.
11. Patient previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody or small molecule tyrosine kinase inhibitor.
12. Patient has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement will not be excluded from the study.
13. Patient has an active infection requiring systemic therapy.
14. Patient has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Patient has a known history of or is positive for Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative] is detected). Patients will be tested for hepatitis B or C infections during screening if they are considered by the investigator to be at higher risk for these infections and have not been previously tested.
16. Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
17. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
19. Patient has received a live vaccine within 30 days prior to first dose.
20. Patient requires concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel).

Allowed anticoagulants are the following:

1. Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.

2. Low-dose low molecular weight heparins (LMWH) are permitted. 3. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor

21. Patient has experienced any of the following within 3 months before the first dose of study treatment:

a. clinically-significant hematemesis, hematuria or gastrointestinal bleeding b. Clinically-significant hemoptysis of > or = 0.5 teaspoon (2.5ml) of red blood c. any other signs indicative of pulmonary hemorrhage

22. Present use or anticipated need for strong CYP3A4 inducers or inhibitors listed below. Patients may not have received a strong CYP3A4 inducer within 12 days prior to registration nor a strong CYP3A4 inhibitor within 7 days prior to registration. Because the lists of these agents are constantly changing, it is important to regularly consult a comprehensive list such as the one located at http://medicine.iupui.edu/clinpharm/ddis/.

* Inducers - dexamethasone; phenytoin; carbamazepine; rifampin; rifabutin; rifapentin; phenobarbital; St. John's Wort
* Inhibitors - Boceprevir; Conivaptan; Indinavir; Itraconazole; Nelfinavir; Ketoconazole; Lopinavir/ritonavir; Mibefradil; Saquinavir; Nefazodone; Telaprevir; Posaconazole; Ritonavir; Voriconazole; Clarithromycin; Telithromycin.

  23. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  a) Cardiovascular disorders including: i) Congestive heart failure (CHF): New York Heart Association (NYHA) Class 3 (moderate) or Class 4 (severe) at the time of screening.

ii) Concurrent uncontrolled hypertension defined as sustained BP > or = 150 mm Hg systolic (grade 2), or > or = 90 mm Hg diastolic (grade 2) despite optimal antihypertensive treatment. (Note: If there is any BP measurement that is performed within the screening period that is < 150 mm Hg systolic and < 90 mm Hg diastolic, then BP does not meet definition of sustained.) iii) Any congenital history of long QT syndrome. iv) Any of the following within 6 months before the first dose of study treatment: v) unstable angina pectoris

* clinically-significant cardiac arrhythmias
* stroke (including TIA, or other ischemic event)
* myocardial infarction
* thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study vi) Cavitating pulmonary lesions(s) or known endotracheal or endobronchial disease manifestation.

vii) Lesions invading or encasing any major blood vessels.

b) Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including: i) Any of the following within 28 days before the first dose of study treatment:

• intra-abdominal tumor/metastases invading GI mucosa (malignant abdominal ascites does not constitute mucosal invasion)

* active peptic ulcer disease,
* inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
* malabsorption syndrome] ii) Any of the following within 6 months before the first dose of study treatment:
* history of abdominal fistula
* gastrointestinal perforation
* bowel obstruction or gastric outlet obstruction
* intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months ago.

iii) GI surgery (particularly when associated with delayed or incomplete healing) within 28 days. Note: Complete healing following abdominal surgery must be confirmed prior to initiating treatment with cabozantinib even if surgery occurred more than 28 days ago.

c) Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea and esophagus.

d) Moderate or severe hepatic impairment.

e) Other clinically significant disorders such as: i) active infection requiring systemic treatment within 28 days before the first dose of study treatment ii) serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment iii) history of organ transplant iv) concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment v) Major surgery (eg, thoracotomy, removal or biopsy of brain metastasis) within 1 month before Week 1 Day 1, minor surgery (eg, simple excision, tooth extraction) at least 10 days before Week 1 Day 1. Subjects with clinically relevant ongoing complications from prior surgery are not eligible. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment.

24. The subject has organ and marrow function and laboratory values as follows:

Hematological:

* Absolute neutrophil count (ANC) < 1,500/mm3/mcL
* White blood cell count < 2,500/mm3
* Platelets < 100,000/mm3/mcL
* Hemoglobin < 9 g/dL- transfusion of packed red blood cells allowed up to 7 days prior to D1.

Renal:

* Serum creatinine > 1.5 X upper limit of normal (ULN), GFR < 30 ml/min
* Serum electrolytes: Serum phosphorus, magnesium, and potassium < LLN after adequate supplementation if necessary

Hepatic:

* Serum total bilirubin > 1.5 X ULN. Patients with a total bilirubin > 1.5 X ULN will not be excluded if Direct bilirubin </= ULN
* AST (SGOT) and ALT (SGPT) > 2.5 X ULN
* Albumin < 2.8 g/dl

Coagulation • International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) > 1.3 X ULN (Patients on oral anticoagulation are excluded.)

Urine

• Urine protein/creatinine ratio (UPCR) > 1 (113.2 mg/mmol) creatinine or 24-hr urine protein of >/= 1 g

25. Cardiovascular: The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >/= 500ms within 14 days before Cycle 1 Day 1. Ejection fraction on Echo or MUGA </= 45%. NYHA class >/= 3. Note: If a single ECG show a QTcF with an absolute value >/= 500 ms, two additional ECGs at intervals of at least 2 minutes must be performed within 30 minutes after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rieth, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Cabozantinib and Pembrolizumab (40mg): Cabozantinib will be administered in the tablet form, at 40 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Cabozantinib: Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form at 40 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Pembrolizumab: Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
- Phase I: Cabozantinib and Pembrolizumab (60mg): Cabozantinib will be administered in the tablet form, at 60 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Cabozantinib: Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form at 60 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Pembrolizumab: Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
- Phase II: Cabozantinib and Pembrolizumab (40 mg): Cabozantinib will be administered in the tablet form at the Recommended Phase 2 dose (RP2D), 40 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Cabozantinib: Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form 40 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Pembrolizumab: Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
Period: Overall Study
Arm/Group | Phase I: Cabozantinib and Pembrolizumab (40mg) | Phase I: Cabozantinib and Pembrolizumab (60mg) | Phase II: Cabozantinib and Pembrolizumab (40 mg)
Started | 6 | 2 | 20
Completed | 1 | 0 | 2
Not Completed | 5 | 2 | 18
Not completed — Adverse Event | 2 | 2 | 6
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Disease progression | 1 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Cabozantinib and Pembrolizumab (40mg); Phase I: Cabozantinib and Pembrolizumab (60mg); Phase II: Cabozantinib and Pembrolizumab: Cabozantinib will be administered in the tablet form, at three dose levels: 40, 20 and 60 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Cabozantinib: Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form, at three dose levels: 40, 20 and 60 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Pembrolizumab: Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
- Total: Total of all reporting groups
Arm/Group | Phase I: Cabozantinib and Pembrolizumab (40mg) | Phase I: Cabozantinib and Pembrolizumab (60mg) | Phase II: Cabozantinib and Pembrolizumab | Total
Number analyzed (Participants) | 6 | 2 | 20 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 14 | 20
  >=65 years | 2 | 0 | 6 | 8
Age, Continuous [Mean (Full Range); unit: years] | 62 [49 to 79] | 54 [54 to 54] | 54 [27 to 80] | 56 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 12
  Male | 2 | 0 | 14 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 20 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 2 | 20 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 20 | 28

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With a Dose Limiting Toxicity (DLT) Using CTCAE, Version 4.03
Description: All adverse events (AEs) will be considered in DLT assessment unless an event is clearly unrelated to trial treatment. The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 will be used.
Time Frame: Up to 21 days
Population: Number of participants enrolled to Phase I cohorts (6 at 40mg and 2 at 60 mg levels)
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Cabozantinib and Pembrolizumab (60mg): Cabozantinib will be administered in the tablet form at 60 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Cabozantinib: Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form at 60 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Pembrolizumab: Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
Arm/Group | Phase I: Cabozantinib and Pembrolizumab (40mg) | Phase I: Cabozantinib and Pembrolizumab (60mg)
Number analyzed (Participants) | 6 | 2
Participants | 1 | 0

2. Primary Outcome: Phase II: Overall Response Rate
Description: The overall response rate (ORR) is the percentage of patients with a complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1). A complete response (CR) is the disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10 mm, and partial response (PR) is a >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Initiation of treatment up to 2 years
Population: Efficacy endpoints (e.g. ORR) were prespecified only for participants enrolled in Phase II.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Cabozantinib and Pembrolizumab: Phase II dose of Cabozantinib and pembrolizumab based on Phase I
Arm/Group | Phase II: Cabozantinib and Pembrolizumab
Number analyzed (Participants) | 20
Participants | 9

3. Secondary Outcome: Disease Control Rate
Description: The disease control rate (DCR) is the percentage of patients with a complete response (CR), partial response (PR) or stable disease (SD) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1). A complete response (CR) is the disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10 mm, partial response (PR) is a >=30% decrease in the sum of the longest diameter of target lesions, and stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Initiation of treatment up to 2 years
Population: Efficacy endpoints (e.g. DCR) were prespecified only for participants enrolled in Phase II.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Cabozantinib and Pembrolizumab: Phase II dose of Cabozantinib and pembrolizumab based on Phase 1
Arm/Group | Phase II: Cabozantinib and Pembrolizumab
Number analyzed (Participants) | 20
Participants | 15

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the time from study treatment initiation to the date of first documentation of disease progression or death due to any cause. Otherwise, patients were censored at date of last radiographic assessment.
Time Frame: Initiation of treatment up to 2 years
Population: Efficacy endpoints (e.g. PFS) were prespecified only for participants enrolled in Phase II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Cabozantinib and Pembrolizumab
Number analyzed (Participants) | 20
months | 6.6 [2.9 to 29.5]

5. Secondary Outcome: Overall Survival at 2 Years
Description: Overall survival (OS) is defined as the time from study treatment initiation to death due to any cause. Patients still alive were censored at the last date known to be alive. Cumulative OS was descriptively summarized over time with the Kaplan-Meier method. The landmark estimate at 2 years and associated 95% confidence interval is reported.
Time Frame: Initiation of treatment up to 2 years
Population: Efficacy endpoints (e.g. OS) were prespecified only for participants enrolled in Phase II.
Measure: Number (95% Confidence Interval); unit: Percent Probability of Survival
Arm/Group | Phase II: Cabozantinib and Pembrolizumab
Number analyzed (Participants) | 20
Percent Probability of Survival | 63 [37 to 80]

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of signing informed consent through 30 days after the last dose of cabozantinib and/or pembrolizumab treatment, up to 2 years.
Groups:
- Phase II: Cabozantinib and Pembrolizumab (40mg): Cabozantinib will be administered in the tablet form, at three dose levels: 40, 20 and 60 mg per day. Pembrolizumab will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks.
  Cabozantinib: Cabozantinib is an oral small molecule potent inhibitor of pro-invasive receptor tyrosine kinases (RTKs).
  Cabozantinib will be administered in the tablet form, at three dose levels: 40, 20 and 60 mg per day, in combination with pembrolizumab. The drug is taken continuously for 21 days or 3 weeks. This period of time is defined as one treatment cycle.
  Pembrolizumab: Pembrolizumab is a humanized antibody which will be administered as an intravenous infusion at a fixed dose of 200 mg once every 3 weeks in combination with cabozantinib.
Arm/Group | Phase I: Cabozantinib and Pembrolizumab (40mg) | Phase I: Cabozantinib and Pembrolizumab (60mg) | Phase II: Cabozantinib and Pembrolizumab (40mg)
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/2 | 10/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/2 | 7/20
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Cabozantinib and Pembrolizumab (40mg) (N=6) | Phase I: Cabozantinib and Pembrolizumab (60mg) (N=2) | Phase II: Cabozantinib and Pembrolizumab (40mg) (N=20)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Cabozantinib and Pembrolizumab (40mg) (N=6) | Phase I: Cabozantinib and Pembrolizumab (60mg) (N=2) | Phase II: Cabozantinib and Pembrolizumab (40mg) (N=20)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 6 (8)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 8 (8)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 6 (9)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 6 (19) | 0 (0) | 10 (19)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (8)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 9 (11)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 4 (7) | 1 (2) | 3 (4)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (5)
Chills (General disorders and administration site conditions) | 1 (1) | 0 (0) | 1 (1)
Death NOS (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders and administration site conditions) | 4 (6) | 1 (1) | 14 (20)
Fever (General disorders and administration site conditions) | 0 (0) | 0 (0) | 3 (3)
Flu like symptoms (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders and administration site conditions) | 1 (1) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders and administration site conditions) | 3 (4) | 0 (0) | 3 (6)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 5 (17) | 2 (7) | 13 (35)
Alkaline phosphatase increased (Investigations) | 3 (3) | 2 (2) | 10 (16)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 2 (7) | 12 (24)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
GGT increased (Investigations) | 2 (3) | 0 (0) | 6 (11)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (4) | 1 (1) | 6 (8)
Neutrophil count decreased (Investigations) | 4 (4) | 0 (0) | 2 (6)
Platelet count decreased (Investigations) | 1 (2) | 2 (2) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight loss (Investigations) | 4 (5) | 0 (0) | 5 (6)
White blood cell decreased (Investigations) | 2 (7) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 6 (7) | 2 (2) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6) | 2 (2) | 8 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 5 (10)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 8 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 5 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (15) | 2 (2) | 13 (25)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 5 (6)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 6 (10)
Proteinuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 5 (6)
Urine discoloration (Renal and urinary disorders) | 6 (8) | 1 (1) | 7 (9)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (10) | 1 (1) | 6 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 2 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 8 (19)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was terminated early due to changes in the treatment of melanoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT03957551/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT03957551/ICF_001.pdf